CLINICAL TRIAL: NCT06827015
Title: The Effect of Laughter Yoga on Anger Levels and Subjective Well-Being in School-Aged Children
Brief Title: Laughter Yoga's Impact on Children's Anger and Well-Being
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Şirin İnanç, Nurse, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024/1224
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Anger Problems; Spiritual Well-being
Keywords: ANGER; LAUGHTER YOGA; SPIRITUAL WELL-BEING; SCHOOL AGE CHILDREN

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to intervention (laughter yoga) and control groups. Intervention effects will be measured at baseline and end.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Students were randomized into groups based on their classes to prevent information leakage, and using Excel-generated randomization, students with high anger scores were assigned equally (1:1 ratio) to Intervention and Delayed groups. Assignment for each student was determined in sealed envelopes, which were opened after the evaluation, implementing blinding by ensuring that neither the students nor the statisticians were aware of the group allocations.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Receiving Laughter Yoga (Experimental): Eight Laughter Yoga Sessions, Each Lasting 40 Minutes, Conducted Twice a Week, for Students with High Anger Levels
  Interventions: Behavioral: Laughter-Based Anger Reduction Program
- Group Without Any Intervention (No Intervention): Participants Receiving No Intervention to Assess Baseline Anger Levels

INTERVENTIONS:
Behavioral: Laughter-Based Anger Reduction Program — This intervention involves structured Laughter Yoga sessions lasting 40 minutes each, conducted twice a week. It specifically targets students with high anger levels. The program combines breathing exercises, playful laughter activities, and relaxation techniques to reduce stress and promote emotional regulation. Unlike other interventions, this program uniquely emphasizes laughter as a tool for managing anger and enhancing overall well-being.
  Arms: Group Receiving Laughter Yoga

SUMMARY:
This study aims to evaluate the effects of laughter yoga on anger levels and mental well-being in schoolchildren. Research indicates that laughter yoga has the potential to reduce stress and improve communication skills. There have been few studies specifically targeting children with high anger levels and low mental well-being. This study focuses on children under stress or with limited social support. Laughter yoga is a fun and effective technique that can be easily integrated into children's daily lives. The study is expected to provide positive contributions to the educational environment and reduce behavioral issues.

DETAILED DESCRIPTION:
This study is a randomized controlled trial aimed at evaluating the effects of laughter yoga on school-aged children's anger levels and mental well-being. The research encompasses a total of 2958 students from two primary schools in Mersin Akdeniz, using 396 fourth-grade students as the sample. Specifically, this research targets children exposed to stress or limited social support, as there are few studies focusing on children with high anger levels and low mental well-being. Children will be assigned to intervention and delay groups based on simple randomization of their anger scores. This process will be conducted branch-based with the assistance of another researcher, and neither participants nor statisticians will have access to group information. The research will collect data in four stages: pre-test, intervention process, post-test, and a follow-up one month later. At each stage, the Emotion Regulation Scale for Children and the Mental Well-Being Questionnaire will be used. Participants will fill in the Mental Well-Being Questionnaire every night before bed during the intervention period, allowing us to evaluate the study's effects. In the long term, it is expected that integrating laughter yoga into children's daily lives in a fun and effective way will provide positive contributions in educational settings and reduce behavioral problems. Research also indicates that laughter yoga has the potential for stress reduction and enhancing communication skills.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 8-11,
* Being a student who regularly attends the school where the study is conducted between February 3 and June 6, when research data is collected,
* Having written consent from a parent/guardian to participate in the study,
* Being willing to participate in the study, and
* Scoring above the median on the Emotion Regulation Scale for Children.

Exclusion Criteria:

* Having a diagnosed health problem that could interfere with laughter exercises (respiratory issues, heart conditions, musculoskeletal problems),
* Having undergone psychological treatment in the last 3 months,
* Currently participating in another psychological support program, and
* Scoring below the median on the Emotion Regulation Scale for Children.
* The criteria for termination of the intervention are not attending two consecutive sessions and non-compliance with the study protocol.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2025-02-28 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-05-05 (Estimated)

PRIMARY OUTCOMES:
Emotion Regulation Scale for Children (ÇDDÖ) | 2 MONTHS
  Emotion Regulation Scale for Children (ÇDDÖ) is designed to assess emotion regulation skills in children aged 8-12. The scale consists of four subscales: Anger (9 items), Excitement (5 items), Fear (8 items), and Sadness (7 items). Each item is rated using a 4-point Likert scale ranging from 1 (does not describe me at all) to 4 (describes me completely). In the reliability and validity study of the Turkish version, the Cronbach's Alpha coefficient was found to be 0.85 for the overall scale. Additionally, there are reverse-scored items (Anger items: 2, 9; Excitement items: 4, 5; Fear items: 3, 6, 7).An increase in the total score indicates an improvement in emotion regulation levels. The average score is 79.50 ± 11.11. Scores below 68.39 indicate poor emotion regulation skills, while scores above 90.61 indicate a positive condition. The ÇDDÖ is planned to be administered on three different occasions: as a pre-test,post-test, and one-month follow-up.
Mental Well-Being Survey | 2 Months
  This survey study aims to evaluate children's daily emotional states using a visual tool. Every day before going to bed, children select the expression that best reflects their emotional state. For evaluation, five facial expressions rated from 1 (very sad) to 5 (very happy) will be used. The scores of the facial expressions selected each day will be collected over a period of 30 days.
  The collected scores will help determine whether a child's mood trends positively or negatively. In the planned study, the minimum score will be 5, and the maximum score will be 25. Based on these scores, values above the average will be considered indicators of a positive mood, while values below the average will be viewed as signs of a negative emotional state.
  The study is planned to include a 4-week measurement and subsequently the first-month measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Emine Öncü, Advisor, Study Director — Mersin University
Locations (2):
- Turkey (Türkiye) (2):
  - Ahmet Mete Işıkara Primary School, Akdeniz, Mersin
  - Hurriyet Primary School, Akdeniz, Mersin

IPD SHARING:
Plan to Share IPD: No
If someone wants to use the data, they will request permission, and it will be shared based on suitability.